CLINICAL TRIAL: NCT04103528
Title: Effects of Procedure Started in the Morning and Afternoon on Early Postoperative Sleep Function and Postoperative Recovery in Patients Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HHT
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Complications
Keywords: Postoperative sleep disturbances; Postoperative recovery; General anesthesia; Early postoperative sleep; Procedure started in the morning and afternoon
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morning group(from 8:00 to 12:00) (Other)
  Interventions: Other: morning surgery
- afternoon group(from 14:00 to 18:00) (Other)
  Interventions: Other: afternoon surgery

INTERVENTIONS:
Other: morning surgery — 31 patients will be operated on between 8:00 and 12:00 in the morning.
  Arms: morning group(from 8:00 to 12:00)
Other: afternoon surgery — 31 patients will be operated on between 14:00 and 18:00 in the afternoon.
  Arms: afternoon group(from 14:00 to 18:00)

SUMMARY:
The present study was conducted in laparoscopic hysteromyoma patients, aiming to compare the effects of morning surgery with afternoon surgery on early postoperative sleep function and postoperative recovery under general anesthesia.

DETAILED DESCRIPTION:
The circadian rhythm is an intrinsic timing mechanism generated by endogenous systems to adapt to the external environment, which is closely related to the human sleep-wake cycle. Patients after major surgery are prone to changes in sleep structure and sleep quality, called postoperative sleep disturbances (POSD), which are characterized by the total sleep time reduced, rapid eye movement sleep absent, slow wave sleep shortened, and shallow sleep phase increased, times of wakefulness increased, and highly fragmented sleep. Some studies have shown that POSD can aggravate postoperative pain and fatigue, increase postoperative delirium, cardiovascular adverse events, and even cause accidental death of patients. The investigators don't know whether the early postoperative sleep function and postoperative recovery quality of patients undergoing general anesthesia are affected by surgery in the morning or in the afternoon. The present study was conducted in laparoscopic hysteromyoma patients, aiming to compare the effects of morning surgery with afternoon surgery on early postoperative sleep function and postoperative recovery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-60 years old.
2. ASA status I or II.
3. BMI 18.5-28 kg/m^2.
4. performed with laparoscopic myomectomy.

Exclusion Criteria:

1. combining with ovarian disease or ovarian surgery.
2. preoperative Athens Insomnia Scale (AIS) score ≥ 4 points
3. chronic use of sedative, hypnotic, psychotropic drugs.
4. recent night shift, cross-time zone, irregular life routine.
5. suffering from mental illness or hearing, visual impairment, and existing sleep apnea syndrome.
6. patients withdraw, or were unable to complete the trial after surgery.
7. lossed bleeding volume more than 500 ml during surgery.
8. performed procedure time exceeded 2 h.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative sleep disturbances by Athens Insomnia Scale | 1 day after the operation
  1. Postoperative sleep disturbances were defined as the total score of Athens Insomnia Scale more than 6.
  2. The incidence of postoperative sleep disturbances was defined as the percentage of the population with a score greater than 6
The sleep time by bispectral index(BIS) monitor from 21:00 to 06:00 on the first night after surgery | 1 day after the operation
  The sleep time: was defined as the total time of BIS values less than 80 during monitoring.
The sleep efficiency by bispectral index(BIS) monitor from 21:00 to 06:00 on the first night after surgery | 1 day after the operation
  The sleep efficiency: was defined as the ratio of a sleeping time over monitoring time.
The sleep quality by bispectral index(BIS) monitor from 21:00 to 06:00 on the first night after surgery | 1 day after the operation
  The sleep quality: was assessed by the area under curve of BIS (BIS-AUC). The BIS-AUC was calculate using the trapezoidal rule, which used trapezium to approximate the region under a curve and calculate its area (GraphPad Prism Version 5.01; San Diego, California). The smaller BIS-AUC was the better sleep quality.

SECONDARY OUTCOMES:
Postoperative recovery Post-operative Quality Recovery Scale(PQRS) | 1 day before surgery (T0), 30 minutes after end of anesthesia (T1), and 1 day after surgery (T2)
  Postoperative Quality Recovery Scale includes five parts: physiological functions (blood pressure, heart rate, temperature, ventilation rate, maintenance of oxygen saturation, airway maintenance, agitation, consciousness, response), Nociceptive (pain, nausea), emotional (depression, anxious), activities of daily living (ability to stand, walk, eat, dress), cognitive function (orientation, digits forward, digits backward, word list, word generation). According to the recovery situation: the physiological function is divided into three levels (3 points: acceptable, 2: abnormality, 1: extreme abnormality), nociceptive, emotional change according to the degree of Likert 5 scored (5: very satisfactory, 4: satisfactory, 3: general, 2: not satisfied, 1: very dissatisfied), and the activities of daily living are equally divided into three levels (3: easy, 2: difficulty, 1: it can't be done completely), when cognitive function score reaches the preoperative baseline level,it means recovery.
The biochemical indicators | 6am one day before and one day after the surgery
  The levels of melatonin (MT), cortisol, and glulcose in the blood were measured separately by ELISA at 6:00am 1 day before and 1 day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan WF, Miao EY, Jin F, Ma H, Lu HW. Changes in First Postoperative Night Bispectral Index After Daytime Sedation Induced by Dexmedetomidine or Midazolam Under Regional Anesthesia: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 May-Jun;41(3):380-6. doi: 10.1097/AAP.0000000000000370. PMID 26928796
- [Result] Brainard J, Gobel M, Bartels K, Scott B, Koeppen M, Eckle T. Circadian rhythms in anesthesia and critical care medicine: potential importance of circadian disruptions. Semin Cardiothorac Vasc Anesth. 2015 Mar;19(1):49-60. doi: 10.1177/1089253214553066. Epub 2014 Oct 7. PMID 25294583
- [Result] Rosenberg-Adamsen S, Kehlet H, Dodds C, Rosenberg J. Postoperative sleep disturbances: mechanisms and clinical implications. Br J Anaesth. 1996 Apr;76(4):552-9. doi: 10.1093/bja/76.4.552. No abstract available. PMID 8652329
- [Result] Hillman DR. Postoperative Sleep Disturbances: Understanding and Emerging Therapies. Adv Anesth. 2017;35(1):1-24. doi: 10.1016/j.aan.2017.07.001. Epub 2017 Sep 18. No abstract available. PMID 29103568
- [Result] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Result] Beydon L, Rauss A, Lofaso F, Liu N, Cherqui D, Goldenberg F, Bonnet F. [Survey of the quality of sleep during the perioperative period. Study of factors predisposing to insomnia]. Ann Fr Anesth Reanim. 1994;13(5):669-74. doi: 10.1016/s0750-7658(05)80723-3. French. PMID 7733516
- [Result] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Result] Su X, Wang DX. Improve postoperative sleep: what can we do? Curr Opin Anaesthesiol. 2018 Feb;31(1):83-88. doi: 10.1097/ACO.0000000000000538. PMID 29120927
- [Result] Gogenur I, Wildschiotz G, Rosenberg J. Circadian distribution of sleep phases after major abdominal surgery. Br J Anaesth. 2008 Jan;100(1):45-9. doi: 10.1093/bja/aem340. Epub 2007 Nov 23. PMID 18037670
- [Result] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Result] Jan JE, Reiter RJ, Wasdell MB, Bax M. The role of the thalamus in sleep, pineal melatonin production, and circadian rhythm sleep disorders. J Pineal Res. 2009 Jan;46(1):1-7. doi: 10.1111/j.1600-079X.2008.00628.x. Epub 2008 Aug 28. PMID 18761566
- [Result] Karkela J, Vakkuri O, Kaukinen S, Huang WQ, Pasanen M. The influence of anaesthesia and surgery on the circadian rhythm of melatonin. Acta Anaesthesiol Scand. 2002 Jan;46(1):30-6. doi: 10.1034/j.1399-6576.2002.460106.x. PMID 11903069
- [Result] de Oliveira Tatsch-Dias M, Levandovski RM, Custodio de Souza IC, Gregianin Rocha M, Magno Fernandes PA, Torres IL, Hidalgo MP, Markus RP, Caumo W. The concept of the immune-pineal axis tested in patients undergoing an abdominal hysterectomy. Neuroimmunomodulation. 2013;20(4):205-12. doi: 10.1159/000347160. Epub 2013 May 8. PMID 23689687
- [Result] Cao M, Javaheri S. Effects of Chronic Opioid Use on Sleep and Wake. Sleep Med Clin. 2018 Jun;13(2):271-281. doi: 10.1016/j.jsmc.2018.02.002. Epub 2018 Mar 12. PMID 29759277
- [Result] Naguib M, Gottumukkala V, Goldstein PA. Melatonin and anesthesia: a clinical perspective. J Pineal Res. 2007 Jan;42(1):12-21. doi: 10.1111/j.1600-079X.2006.00384.x. PMID 17198534
- [Result] Mihara T, Kikuchi T, Kamiya Y, Koga M, Uchimoto K, Kurahashi K, Goto T. Day or night administration of ketamine and pentobarbital differentially affect circadian rhythms of pineal melatonin secretion and locomotor activity in rats. Anesth Analg. 2012 Oct;115(4):805-13. doi: 10.1213/ANE.0b013e3182632bcb. Epub 2012 Aug 10. PMID 22886841
- [Result] Li CX, An XX, Zhao B, Wu SJ, Xie GH, Fang XM. Impact of operation timing on post-operative infections following colorectal cancer surgery. ANZ J Surg. 2016 Apr;86(4):294-8. doi: 10.1111/ans.13471. Epub 2016 Feb 17. PMID 26887845
- [Result] Gimenez S, Romero S, Alonso JF, Mananas MA, Pujol A, Baxarias P, Antonijoan RM. Monitoring sleep depth: analysis of bispectral index (BIS) based on polysomnographic recordings and sleep deprivation. J Clin Monit Comput. 2017 Feb;31(1):103-110. doi: 10.1007/s10877-015-9805-5. Epub 2015 Nov 14. PMID 26578097
- [Result] Dolan R, Huh J, Tiwari N, Sproat T, Camilleri-Brennan J. A prospective analysis of sleep deprivation and disturbance in surgical patients. Ann Med Surg (Lond). 2016 Jan 6;6:1-5. doi: 10.1016/j.amsu.2015.12.046. eCollection 2016 Mar. PMID 26909151
- [Result] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. J Psychosom Res. 2000 Jun;48(6):555-60. doi: 10.1016/s0022-3999(00)00095-7. PMID 11033374
- [Derived] Hou H, Wu S, Qiu Y, Song F, Deng L. The effects of morning/afternoon surgeries on the early postoperative sleep quality of patients undergoing general anesthesia. BMC Anesthesiol. 2022 Sep 10;22(1):286. doi: 10.1186/s12871-022-01828-w. PMID 36088298